CLINICAL TRIAL: NCT00131339
Title: Placebo-Controlled Evaluation of the Efficacy of D-Cycloserine for Enhancing the Effects of CBT for Panic Disorder
Brief Title: Augmenting Exposure Therapy With an N-Methyl-D-Aspartate (NMDA) Agonist for Panic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TOLI001428HI
Record Dates: First submitted 2005-08-16; First posted 2005-08-18 (Estimated); Last update posted 2009-08-26 (Estimated); Status verified 2009-08

CONDITIONS: Panic Disorder
Keywords: panic disorder; cognitive behavioral therapy; D-cycloserine; medication; treatment trial; placebo-controlled; double-blind; randomized
MeSH Terms: conditions — Panic Disorder | interventions — Cognitive Behavioral Therapy; Cycloserine

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy
Drug: D-cycloserine

SUMMARY:
This study involves cognitive behavioral therapy (CBT) and a medication called D-cycloserine (DCS), which is thought to help reduce panic symptoms more effectively by interacting with N-methyl-D-aspartate (NMDA) glutamate receptors, facilitating many forms of learning including the extinction of fear. Participants will be randomly assigned (like flipping a coin) to receive either DCS or a placebo in addition to CBT.

DETAILED DESCRIPTION:
This study consists of cognitive behavioral therapy (CBT) including exposure to physical sensations and feared situations, which have been demonstrated to be effective for many individuals with panic disorder.

All assessments and treatment sessions are free of charge. Half of the patients will be randomly assigned to receive D-cycloserine (DCS) and half wll be assigned to receive a placebo. Although DCS is used in humans to treat tuberculosis, it has not been FDA approved for this indication. Recent research in other anxiety disorders has shown that DCS plus behavior therapy is more effective than behavior therapy alone.

This treatment study had two active interventions. All patients will receive CBT and the researchers expect that everybody will improve from this treatment. However, it may be that those patients in the DCS intervention will improve somewhat more than those in the placebo intervention.

The treatment will be structured with at home practice and repeated assessments. Assessments are extremely important as they guide the treatment and provide the study investigators necessary information about the treatment. The treatment consists of 5 sessions (once a week) plus a one week post-treatment assessment and follow-up assessments at one month and six months.

ELIGIBILITY:
Inclusion Criteria:

* Principal diagnosis of panic disorder

Exclusion Criteria:

* History of psychotic disorders or bipolar disorder
* Substance dependence
* Pregnant or breastfeeding
* History of a medical condition that may increase the risks of taking the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-11; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
significant reduction in panic symptoms after completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael W. Otto, Ph.D., Principal Investigator — Center for Anxiety and Related Disorders at Boston University
Locations (2):
- United States (2):
  - Hartford Hospital, Hartford, Connecticut
  - Center for Anxiety and Related Disorders at Boston University, Boston, Massachusetts

REFERENCES:
- [Derived] Otto MW, Tolin DF, Simon NM, Pearlson GD, Basden S, Meunier SA, Hofmann SG, Eisenmenger K, Krystal JH, Pollack MH. Efficacy of d-cycloserine for enhancing response to cognitive-behavior therapy for panic disorder. Biol Psychiatry. 2010 Feb 15;67(4):365-70. doi: 10.1016/j.biopsych.2009.07.036. Epub 2009 Oct 6. PMID 19811776